CLINICAL TRIAL: NCT02128529
Title: A Cross-sectional Observational Study in Pulmonology Departments in Belgium and Luxembourg to Investigate the Epidemiology of Chronic Bronchitis in Patients Suffering From Moderate to Very Severe COPD
Brief Title: Epidemiology of Chronic Bronchitis in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: RO-2455-401-BE
Record Dates: First submitted 2014-04-29; First posted 2014-05-01 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Obstructive Pulmonary Disease; Chronic Bronchitis
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic obstructive pulmonary disease: Patients with chronic obstructive pulmonary disease will undergo a single visit with the collection of data from his/her records.

SUMMARY:
The purpose of this study was to investigate the prevalence of chronic bronchitis in patients suffering from moderate to very severe chronic obstructive pulmonary disease (COPD), and to assess the difference in exacerbation rates in patients suffering from moderate to very severe COPD with chronic bronchitis vs. a population of patients without chronic bronchitis.

DETAILED DESCRIPTION:
This was an observational study so participants only took medication that was prescribed by their regular healthcare provider. No additional study medication was administered. This study enrolled patients who were previously diagnosed with moderate to very severe chronic obstructive pulmonary disease (COPD). This study looked at the prevalence of chronic bronchitis in patients suffering from moderate, severe or very severe COPD, and it also compared worsening of COPD in patients with or without chronic bronchitis. This study enrolled 976 patients. This multi-centre trial was conducted in Belgium and Luxembourg. The overall time to participate in this study was at a single, regularly scheduled visit at the pulmonologists office. There were no follow-up assessments for this study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Written informed consent. 2. Age ≥ 40 years. 3. Forced expiratory volume in one second (FEV1)/Forced vital capacity (FVC) ratio (post-bronchodilator) <70%. 4. FEV1 (post-bronchodilator) < 80% of predicted.

Exclusion Criteria:

* 1. Moderate and severe exacerbations during the last 4 weeks. 2. Pregnancy. 3. Already participated in the study (allowed to participate only once).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients with or without chronic bronchitis in Belgium and Luxembourg.
Sampling Method: Non-Probability Sample
Enrollment: 976 (Actual)
Dates: Start 2010-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Chronic Bronchitis | 2 years prior to the study visit on Day 1
  Chronic bronchitis is defined as the presence of cough and sputum production for at least 3 months in each of 2 consecutive years.
Exacerbation Rate | 12 Months prior to the study visit
  An exacerbation is defined as an event in the natural course of the disease characterised by a change in the patient's baseline dyspnoea, cough, and/or sputum that is beyond normal day-to-day variations, is acute in onset, and may warrant a change in regular medication in a patient with underlying COPD for three or more days. Exacerbation rate is defined as number of exacerbations per year.

SECONDARY OUTCOMES:
Percentage of Participants with Moderate, Severe or Very Severe COPD | At the study visit (Day 1)
  COPD severity will be assessed based on post-bronchodilator forced expiratory volume after 1 second (FEV1) and post-bronchodilator ratio of FEV1 to forced vital capacity (FVC) and then classified by the Global Initiative for Chronic Obstructive Lung Disease (GOLD): Moderate - FEV1/FVC<0.7, FEV1 50-79% normal; Severe - FEV1/FVC<0.70, FEV1 30-49% normal; Very Severe - FEV1/FVC<0.70, FEV1 <30% predicted or FEV1<50% predicted plus chronic respiratory failure.
Percentage of Participants with Risk Factors | 12 months prior to study visit
  Risk factors are defined as smoking status and exposure to environmental risk factors (mineral dusts, organic dusts, fumes and vapours or metallic dusts).
Changes in Post-bronchodilator forced expiratory volume after 1 second (FEV1) | At the study visit, and 6 months and 12 Months prior to study visit
Percentage of Participants with Other Relevant Diseases | 12 months prior to study visit
  Relevant disease are defined as respiratory diseases (allergy, asthma, chronic respiratory failure), cardiovascular diseases (ischaemic heart disease, heart failure, hypertension), and other diseases (which could be related to COPD) (osteoporosis, skeletal muscle wasting, cachexia, diabetes mellitus, depression, normocytic, anaemia, gastroesophageal reflux disease and lung cancer).
COPD Treatment | At the study visit (Day 1)
  COPD treatments are defined as inhaled therapies, oral therapies and other therapies administered within the last 12 months as influenza vaccination and smoking cessation therapy.
Changes in post-bronchodilator ratio of FEV1 to forced vital capacity (FVC) | At the study visit, and 6 months and 12 Months prior to study visit

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca

REFERENCES:
- See also: Full publication — http://onlinelibrary.wiley.com/doi/10.1111/ijcp.12248/full